CLINICAL TRIAL: NCT01304888
Title: Evaluating the Impact of the Programa de Apoyo Alimentaria
Brief Title: Evaluating the Impact of the Food Support Program (Programa de Apoyo Alimentaria)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Secretaría de Desarrollo Social (SEDESOL) (Unknown)
Responsible Party: Researcher, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: INSP01
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2011-02

CONDITIONS: Malnutrition
Keywords: Food consumption
MeSH Terms: conditions — Malnutrition | interventions — CASP8 and FADD-Like Apoptosis Regulating Protein; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Food basket w/o nutrition education (Experimental)
  Interventions: Other: Food basket w/o nutrition education
- Food basket + nutrition education (Experimental)
  Interventions: Other: Food basket + nutrition education
- Control (Experimental)
  Interventions: Other: Control
- Cash + health and nutrition education (Experimental)
  Interventions: Other: Cash + nutrition education

INTERVENTIONS:
Other: Cash + nutrition education — Cash transfer of 150 Mexican pesos (equivalent to approximately 14 USD at the time) per month. The size of the cash transfer and the amount of food was the same for all households, i.e. no adjustments for family size or composition were made. Households received the transfer once every 2 mo. Beneficiary households were required to attend nutrition and health education sessions and had to participate in program related logistic activities in order to receive the benefits. These program conditionalities, however, were not strictly enforced.
  Arms: Cash + health and nutrition education
Other: Food basket + nutrition education — Monthly food basket with a cost to the program of 150 pesos. The amount of food was the same for all households, i.e. no adjustments for family size or composition were made. The basket contained a number of staple and basic food products and powdered whole milk (Liconsa), which is fortified with Zn, Fe, Vitamin C, and folate. The composition of the food basket conformed to the Mexican norm for food aid programs (NOM-169-SSA1-1998). Households received the transfer once every 2 mo. Beneficiary households were required to attend nutrition and health education sessions and had to participate in program related logistic activities in order to receive the benefits. These program conditionalities, however, were not strictly enforced.
  Arms: Food basket + nutrition education
Other: Food basket w/o nutrition education — A monthly food basket with a cost to the program of 150 pesos. The amount of food was the same for all households, i.e. no adjustments for family size or composition were made. The basket contained a number of staple and basic food products and powdered whole milk (Liconsa), which is fortified with Zn, Fe, Vitamin C, and folate. The composition of the food basket conformed to the Mexican norm for food aid programs (NOM-169-SSA1-1998). Households received the transfer once every 2 mo. Beneficiary households were not required to attend nutrition and health education sessions.
  Arms: Food basket w/o nutrition education
Other: Control — No benefits were provided
  Arms: Control

SUMMARY:
The Programa de Apoyo Alimentaria (PAL) started in 2003 and is targeted to communities in Mexico that do not receive benefits from other federal food aid programs, have less than 2,500 inhabitants and a high level of marginalization. Marginalization is a term used in Mexico for the multidimensional assessment of poverty in a community.

When the program started in 2003 it provided beneficiary households either a cash transfer of 150 Mexican pesos (equivalent to approximately 14 USD at the time) per month or a monthly food basket with a cost to the program of 150 pesos. The size of the cash transfer and the amount of food was the same for all households, i.e. no adjustments for family size or composition were made. The basket contained a number of staple and basic food products and powdered whole milk (Liconsa), which is fortified with Zn, Fe, Vitamin C, and folate (Table 1). The composition of the food basket conformed to the Mexican norm for food aid programs (NOM-169-SSA1-1998), which states that food transfers need to provide at least 20% of the recommended daily energy and protein requirements. Beneficiary households were required to attend nutrition and health education sessions and had to participate in program related logistic activities in order to receive the benefits. These program conditionalities, however, were not strictly enforced.

A community randomized controlled intervention trial was used to evaluate the impact of the intervention. A random sample of 208 rural communities was drawn from the pool of eligible communities in 8 of the poorest states in the South/Eastern region of Mexico (Chiapas, Guerrero, Oaxaca, Quintana Roo, Tabasco, Campeche, Yucatan and Veracruz). Within each community a random sample of 33 households was selected. The baseline survey was conducted from October 2003 to April 2004. After baseline data collection, the 208 selected communities (6,687 households) randomly assigned to one of four study groups: food basket without education (52 communities, 1657 households), food basket with education (52 communities, 1680 households), cash transfer with education (53 communities, 1687 communities) or control (51 communities, 1663 households). Treatment allocation was carried out by the Ministry of Social Development.

ELIGIBILITY:
Inclusion Criteria:

* Live in a community that does not receive benefits from other federal food aid programs, have less than 2,500 inhabitants and a high level of marginalization. Marginalization is a term used in Mexico for the multidimensional assessment of poverty in a community. It takes into account housing quality (including the percent of households without piped water, without sewage and without electricity), income (proportion of household below two times the minimum wage), education (including illiteracy) and urbanization.
* Households within these communities were eligible if they fell below the "needs" poverty line as defined by the Mexican Ministry of Social Development. This corresponds to an income level sufficient to cover basic needs in food consumption, health and education.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6687 (Actual)
Dates: Start 2003-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Child nutritional status

SECONDARY OUTCOMES:
Household food consumption

OTHER OUTCOMES:
Body weight

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Gonzalez de Cossio, PhD, Principal Investigator — National Institute of public Health
Locations (1):
- Instituto Nacional de Salud Publica, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Result] Leroy JL, Gadsden P, Rodriguez-Ramirez S, de Cossio TG. Cash and in-kind transfers in poor rural communities in Mexico increase household fruit, vegetable, and micronutrient consumption but also lead to excess energy consumption. J Nutr. 2010 Mar;140(3):612-7. doi: 10.3945/jn.109.116285. Epub 2010 Jan 20. PMID 20089777
- [Derived] Ramirez-Luzuriaga MJ, Unar-Munguia M, Rodriguez-Ramirez S, Rivera JA, Gonzalez de Cosio T. A Food Transfer Program without a Formal Education Component Modifies Complementary Feeding Practices in Poor Rural Mexican Communities. J Nutr. 2016 Jan;146(1):107-13. doi: 10.3945/jn.115.215962. Epub 2015 Nov 11. PMID 26561408